CLINICAL TRIAL: NCT02683577
Title: A Phase 1, Open-label Study to Evaluate the Single Dose Pharmacokinetics of Telotristat Etiprate in Male and Female Subjects With Mild, Moderate and Severe Hepatic Impairment and Matched Subjects With Normal Hepatic Function
Brief Title: Study to Evaluate a Dose of Telotristat Etiprate in Male and Female With Mild, Moderate and Severe Hepatic Insufficiency and Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D-FR-01017-001; 2015-004120-64 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — telotristat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telotristat etiprate 500 mg (Experimental): 1 single oral dose (2 x 250-mg tablets)
  Interventions: Drug: telotristat etiprate

INTERVENTIONS:
Drug: telotristat etiprate

SUMMARY:
The purpose of the protocol is to assess the pharmacokinetics, safety and tolerability of a single dose of telotristat etiprate in subjects with various stages of hepatic impairment compared to healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 34 kg/m², inclusive, at screening. BMI 35 may be accepted in case of 3-point scored ascites.
* Minimum body weight of 50 kg.
* Vital signs (after 5 minutes resting in a supine position) that are within study specified ranges
* Female subjects of childbearing potential must agree to use an adequate double-barrier method of contraception during the study and for 30 days after discharge.
* Subjects with impaired hepatic function: Clinical diagnosis of chronic hepatic disease (stable for more than 3 months) with a documented history of underlying hepatic insufficiency and no acute episodes of illness within 30 days prior to Day -1, and no significant change in disease status (ie, up to 1 point in the Child-Pugh classification) from screening to Day -1.
* Control subjects with normal hepatic function: Clinical laboratory test results must be strictly within the normal laboratory reference ranges for liver function, and mean corpuscular volume (MCV) or, for other parameters, deemed as not clinically significant by the investigator.

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or Electrocardiogram (ECG) findings (with the exception of those parameters that are resulting from the underlying hepatic disease) that, in the opinion of the investigator, may interfere with any aspect of study conduct or interpretation of results.
* Clinically significant illness or disease as determined by medical history, including cardiac, pulmonary, hepatic (other than reason for their hepatic impairment), biliary, Gastrointestinal (GI), endocrinologic, or renal disorders, or cancer within the last 5 years (except localised or in situ nonmelanoma skin cancer), physical examination, clinical laboratory tests, and 12-lead ECGs.
* Receipt of any investigational agent or study drug within 30 days or 10 half-lives, whichever is longer, prior to dosing.
* Smoking more than 20 cigarettes (eg, 1 pack) per day or equivalent (eg, e-vapour cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum); unable or unwilling to refrain from smoking and tobacco use for 2 hours prior to dosing and 4 hours after dose administration.
* History of any serious adverse reaction or hypersensitivity to any inactive component of telotristat etiprate (ie, microcrystalline cellulose, croscarmellose sodium (disintegrant), talc, silicon dioxide, and magnesium stearate (nonbovine)).
* Existence of any surgical or medical condition that, in the judgment of the investigator and the sponsor's, medical monitor, might interfere with the absorption, distribution, metabolism, or excretion of telotristat etiprate.
* History of any major surgery within 6 months or anticipated surgery prior to Day -1.
* History of renal disease or significantly abnormal kidney function test.
* History of any active infection within 30 days prior to Day 1, if deemed clinically significant by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- ARENSIA Exploratory Medicine, Chisinau, Moldova
- ARENSIA Exploratory Medicine, Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study conducted at 2 investigational sites, one in Romania and one in the Republic of Moldova. Subjects were enrolled to the study from 08 February 2016 (first subject enrolled) until 07 July 2016 (last subject completed).
Pre-assignment Details: Subjects enrolled into 3 hepatic functional groups:
  * Healthy control subjects with normal hepatic function
  * Mild hepatic impairment (HI) subjects (Child-Pugh [C-P] class A)
  * Moderate HI subjects (C-P class B).
  C-P score was summed from 5 clinical assessments of liver disease; each measure scored 1-3, with 3 indicating most severe derangement.
Groups:
- Healthy Control: Subjects in the healthy control group were assessed as having normal hepatic function.
  All subjects in each study group received a single oral dose of telotristat ethyl hippurate 500 mg (2x250 mg) on Day 1.
- Mild HI: Subjects in the mild HI group were assessed as C-P class A (5 to 6 points on C-P scale for classification of the severity of liver disease).
  All subjects in each study group received a single oral dose of telotristat ethyl hippurate 500 mg (2x250 mg) on Day 1.
- Moderate HI: Subjects in the moderate HI group were assessed as C-P class B (7 to 9 points on C-P scale for classification of the severity of liver disease).
  All subjects in each study group received a single oral dose of telotristat ethyl hippurate 500 mg (2x250 mg) on Day 1.
Period: Overall Study
Arm/Group | Healthy Control | Mild HI | Moderate HI
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the safety population which corresponds to all subjects who received at least one dose of study medication.
Arm/Group | Healthy Control | Mild HI | Moderate HI | Total Title
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 7 | 22
  >=65 years | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 5 | 4 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Maximum Observed Plasma Drug Concentration (Cmax) for Telotristat Ethyl and Comparison Between Each HI Group and Healthy Control Group
Description: Blood was sampled for the purpose of determining pharmacokinetic (PK) parameters for total telotristat ethyl using a validated, specific, and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) bioanalytical method. The method was selective, linear, precise and accurate within the range from 0.5 to 500 nanograms per millilitre (ng/mL) for telotristat ethyl and the lower limit of quantification (LoQ) was 0.5 ng/mL. Results were derived by non-compartmental analysis of the plasma concentration-time profiles.
Time Frame: Blood samples were collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours [h] post-dose), Day 2 (24 h), Day 3 (48 h) and Day 4 (72 h).
Population: The PK population (23 subjects overall) corresponded to all subjects who received at least one dose of study medication, without protocol violation affecting PK evaluation and who had a sufficient number of plasma concentrations to estimate the main PK parameters (Cmax, Tmax and AUC[0-tlast]).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- All HI: The all HI group represented all subjects in either HI group (mild + moderate). All subjects in each study group received a single oral dose of telotristat ethyl hippurate 500 mg (2x250 mg) on Day 1.
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
ng/mL | 4.06 (54.4) | 6.88 (106.6) | 9.99 (47.8) | 8.19 (81.0)
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; Comparison of mild HI group (Test) versus healthy control group (Reference) for Cmax values for telotristat ethyl; Test type: Superiority or Other; Geometric least square (LS) mean ratio = 1.695, 90% CI 2-sided [0.904 to 3.176] — A repeated-measures analysis of variance (ANOVA) was performed using a linear mixed effects model, with hepatic function group as a fixed term. Geometric LS mean ratios were derived for each HI group (Test) versus healthy control group (Reference)
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; Comparison of moderate HI group (Test) versus healthy control group (Reference) for Cmax values for telotristat ethyl; Test type: Superiority or Other; Geometric LS mean ratio = 2.462, 90% CI 2-sided [1.579 to 3.837] — A repeated-measures ANOVA was performed using a linear mixed effects model, with hepatic function group as a fixed term. Geometric LS mean ratios were derived for each HI group (Test) versus healthy control group (Reference)

2. Primary Outcome: Assessment of Time to Maximum Observed Plasma Concentration (Tmax) for Telotristat Ethyl and Comparison Between Each HI Group and Healthy Control Group
Description: Blood was sampled for the purpose of determining PK parameters for total telotristat ethyl using a LC-MS/MS bioanalytical method. The method was selective, linear, precise and accurate within the range from 0.5 to 500 ng/mL for telotristat ethyl and the LoQ was 0.5 ng/mL. Results were derived by non-compartmental analysis of the plasma concentration-time profiles.
Time Frame: Blood samples were collected on Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 h post-dose), Day 2 (24 h), Day 3 (48 h) and Day 4 (72 h).
Population: The PK population corresponded to all subjects who received at least one dose of study medication, without protocol violation affecting PK evaluation and who had a sufficient number of plasma concentrations to estimate the main PK parameters (Cmax, Tmax and AUC[0-tlast]).
Measure: Median (Full Range); unit: hour
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
hour | 1.000 [0.50 to 3.00] | 1.000 [0.50 to 3.00] | 1.000 [0.50 to 1.00] | 1.000 [0.50 to 3.00]
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; The Tmax was analysed using a non-parametric analysis (Walsh averages and appropriate quantile of the Wilcoxon signed rank test statistic). The median difference between the mild HI group (Test) versus healthy control group (Reference) and the corresponding 90% CIs were calculated by Hodges-Lehmann estimation; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney); Median difference = 0.000, 90% CI 2-sided [0.000 to 0.000]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; The Tmax was analysed using a non-parametric analysis (Walsh averages and appropriate quantile of the Wilcoxon signed rank test statistic). The median difference between the moderate HI group (Test) versus healthy control group (Reference) and the corresponding 90% CIs were calculated by Hodges-Lehmann estimation; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney); Median difference = 0.000, 90% CI 2-sided [0.000 to 0.000]

3. Primary Outcome: Assessment of Area Under the Plasma Concentration Time Curve From 0 to Time t Corresponding to the Last Quantifiable Concentration (AUC[0-tlast]) for Telotristat Ethyl and Comparison Between Each HI Group and Healthy Control Group
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
ng*h/mL | 4.94 (85.5) | 11.33 (100.5) | 15.65 (62.7) | 13.17 (82.5)
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; Comparison of mild HI group (Test) versus healthy control group (Reference) for AUC(0-tlast) values for telotristat ethyl; Test type: Superiority or Other; Geometric LS mean ratio = 2.294, 90% CI 2-sided [1.144 to 4.598] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; Comparison of moderate HI group (Test) versus healthy control group (Reference) on AUC(0-tlast) values for telotristat ethyl; Test type: Superiority or Other; Geometric LS mean ratio = 3.168, 90% CI 2-sided [1.715 to 5.852] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Assessment of Area Under the Plasma Concentration Time Curve From Time 0 to Infinity (AUC[0-inf]) for Telotristat Ethyl
Description: Blood was sampled for the purpose of determining PK parameters for total telotristat ethyl using a LC-MS/MS bioanalytical method. The method was selective, linear, precise and accurate within the range from 0.5 to 500 ng/mL for telotristat ethyl and the LoQ was 0.5 ng/mL. Results were derived by non-compartmental analysis of the plasma concentration-time profiles. AUC(0-inf) was not determined when the apparent terminal elimination half-life (t1/2) could not be determined over a time interval equal to at least 2 times t1/2 and/or the adjusted coefficient of determination value was inferior to 0.7 and/or extrapolated AUC was greater than 20%.
Time Frame: as for outcome 2
Population: The PK population corresponded to all subjects who received at least one dose of study medication, without protocol violation affecting PK evaluation and who had a sufficient number of plasma concentrations to estimate the main PK parameters (Cmax, Tmax and AUC[0-tlast]). Only subjects with data available for analysis are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 3 | 7 | 6 | 13
ng*h/mL | NA (NA) — No descriptive statistics were computed when more than 1/3 of the PK parameter values were not determined. | 11.70 (108.4) | 17.79 (58.5) | 14.20 (86.5)

5. Primary Outcome: Assessment of Cmax for LP-778902 (Active Metabolite) and Comparison Between Each HI Group and Healthy Control Group
Description: Blood was sampled for the purpose of determining PK parameters for LP-778902 (active metabolite of telotristat ethyl) using a LC-MS/MS bioanalytical method. The method was selective, linear, precise and accurate within the range from 2 to 2000 ng/mL for LP-778902 and the LoQ was 2.0 ng/mL. Results were derived by non-compartmental analysis of the plasma concentration-time profiles.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
ng/mL | 666.1 (36.4) | 1143.9 (65.7) | 1333.3 (25.2) | 1228.7 (48.6)
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; Comparison of mild HI group (Test) versus healthy control group (Reference) for Cmax values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 1.72, 90% CI 2-sided [1.11 to 2.65] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; Comparison of moderate HI group (Test) versus healthy control group (Reference) on Cmax values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 2.00, 90% CI 2-sided [1.51 to 2.66] — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Assessment of Tmax for LP-778902 (Active Metabolite) and Comparison Between Each Hepatic Impairment Group and Healthy Control Group and Comparison Between Each Hepatic Impairment Group and Healthy Control Group
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
hour | 2.000 [1.00 to 3.00] | 2.000 [2.00 to 3.00] | 2.000 [2.00 to 3.00] | 2.000 [2.00 to 3.00]
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; The Tmax was analysed using a non-parametric analysis (Walsh averages and appropriate quantile of the Wilcoxon signed rank test statistic). The median differences between the hepatic impaired group (Test) versus the healthy control group (Reference) and the corresponding 90% CIs were calculated by Hodges-Lehmann estimation; Test type: Superiority or Other; p = 0.3160, Wilcoxon (Mann-Whitney); Median difference = 0.000, 90% CI 2-sided [0.000 to 1.000]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.4671, Wilcoxon (Mann-Whitney); Median difference = 0.000, 90% CI 2-sided [0.000 to 1.000]

7. Primary Outcome: Assessment of AUC(0-tlast) for LP-778902 (Active Metabolite) and Comparison Between Each Hepatic Impairment Group and Healthy Control Group
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 8 | 8 | 7 | 15
ng*h/mL | 2436.5 (36.3) | 5831.2 (82.6) | 8565.4 (45.5) | 6977.2 (68.0)
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; Comparison of mild HI group (Test) versus healthy control group (Reference) on AUC(0-tlast) values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 2.39, 90% CI 2-sided [1.45 to 3.94] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; Comparison of moderate HI group (Test) versus healthy control group (Reference) on AUC(0-tlast) values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 3.52, 90% CI 2-sided [2.45 to 5.03] — [estimate comment as in outcome 1, analysis 2]

8. Primary Outcome: Assessment of AUC(0-inf) for LP-778902 (Active Metabolite) and Comparison Between Each HI Group and Healthy Control Group
Description: Blood was sampled for the purpose of determining PK parameters for LP-778902 (active metabolite of telotristat ethyl) using a LC-MS/MS bioanalytical method. The method was selective, linear, precise and accurate within the range from 2 to 2000 ng/mL for LP-778902 and the LoQ was 2.0 ng/mL. Results were derived by non-compartmental analysis of the plasma concentration-time profiles. AUC(0-inf) was not determined when terminal half-life (t1/2) could not be determined over a time interval equal to at least 2 times t1/2 and/or the adjusted coefficient of determination value was inferior to 0.7 and/or extrapolated AUC was greater than 20%.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 7 | 8 | 7 | 15
ng*h/mL | 2599.0 (34.2) | 5866.5 (82.3) | 8626.3 (45.7) | 7022.9 (67.9)
Statistical Analysis 1: Comparison: Healthy Control vs Mild HI; Comparison of mild HI group (Test) versus healthy control group (Reference) on ln transformed AUC(0-inf) values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 2.26, 90% CI 2-sided [1.33 to 3.82] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Healthy Control vs Moderate HI; Comparison of moderate HI group (Test) versus healthy control group (Reference) on AUC(0-inf) values for LP-778902; Test type: Superiority or Other; Geometric LS mean ratio = 3.32, 90% CI 2-sided [2.30 to 4.80] — [estimate comment as in outcome 1, analysis 2]

9. Primary Outcome: Assessment of t1/2 for Telotristat Ethyl and LP-778902 (Active Metabolite)
Description: Blood was sampled for the purpose of determining PK parameters for total telotristat ethyl and its active metabolite LP-778902 using a LC-MS/MS bioanalytical method. The method was selective, linear, precise and accurate within the range from 0.5 to 500 ng/mL for telotristat ethyl and from 2 to 2000 ng/mL for LP-778902. The LoQ for telotristat ethyl and its metabolite LP-778902 were 0.5 ng/mL and 2.0 ng/mL, respectively.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 7 | 8 | 7 | 15
hour
  Telotristat ethyl: number analyzed (Participants) | 3 | 7 | 6 | 13
  Telotristat ethyl | NA (NA) — No descriptive statistics were computed when more than 1/3 of the PK parameter values were not determined. | 0.901 (31.1) | 1.002 (31.2) | 0.947 (30.3)
  LP-778902 | 9.12 (6.8) | 10.96 (12.7) | 11.08 (10.8) | 11.02 (11.5)

10. Primary Outcome: Assessment of Apparent Terminal Elimination Rate Constant (λz) for Telotristat Ethyl and LP-778902 (Active Metabolite)
Description: as for outcome 9
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour^-1
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Number analyzed (Participants) | 7 | 8 | 7 | 15
hour^-1
  Telotristat ethyl: number analyzed (Participants) | 3 | 7 | 6 | 13
  Telotristat ethyl | NA (NA) — No descriptive statistics were computed when more than 1/3 of the PK parameter values were not determined. | 0.769 (31.1) | 0.691 (31.2) | 0.732 (30.3)
  LP-778902 | 0.08 (6.8) | 0.06 (12.7) | 0.06 (10.8) | 0.06 (11.5)

ADVERSE EVENTS:
Time Frame: Up to 15 days (Day 1 to Day 15)
Description: Adverse event (AE) data is reported for the safety population which corresponds to all subjects who received at least one dose of study medication (24 subjects overall). Data is reported as treatment-emergent AEs, defined as any AE occurring during the active phase of the study until the end of study or early discontinuation visit.
Arm/Group | Healthy Control | Mild HI | Moderate HI | All HI
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 3/8 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control (N=8) | Mild HI (N=8) | Moderate HI (N=8) | All HI (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
No safety risks were identified in mild or moderate HI subjects but due to uncertainties regarding potential exposure of study medication in severe HI subjects, it was decided not to enrol any subjects with severe HI (optional as per the protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide the sponsor with any results communications for public release at least 90 days prior to the planned submission for their review.